CLINICAL TRIAL: NCT01986582
Title: Stage 2, Double-blind, Randomized, Parallel Groups, One Centre Study in Patients With Allergic Rhinitis Treated With Nasal Oxymetazoline in Combination With Nasal Hydroxyl-propyl-methyl Cellulose (HPMC) or Placebo
Brief Title: NoAL (HPMC) in Combination With Oxymetazoline in Patients With Allergic Rhinitis
Acronym: NOPAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association Asthma, Bulgaria (Other)
Collaborators: Nasaleze (Industry)
Responsible Party: Principal Investigator, Prof. Todor Popov, Professor, Association Asthma, Bulgaria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NoAL001
Record Dates: First submitted 2013-11-12; First posted 2013-11-18 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Congestion; Mucoadhesive Treatment; Nasal Decongestant
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): One puff of oxymetazoline immediately followed by one puff of hydroxyl-propyl-methyl cellulose powder, morning & evening, for 8 days.
  Interventions: Drug: Oxymetazoline; Other: Hydroxyl-propyl-methyl cellulose powder
- Group B (Placebo Comparator): One puff of oxymetazoline immediately followed by one puff of placebo, morning & evening, for 8 days.
  Interventions: Drug: Oxymetazoline; Other: Placebo (lactose powder)

INTERVENTIONS:
Drug: Oxymetazoline — Intranasal application
  Other Names: Afrin
Other: Hydroxyl-propyl-methyl cellulose powder — Intranasal application
  Other Names: NoAl
  Arms: Group A
Other: Placebo (lactose powder) — Intranasal application
  Arms: Group B

SUMMARY:
Allergic rhinitis is treated with a variety of systemic and locally applied drugs. The effectiveness of the intranasally applied formulations is diminished by the cleaning mechanisms of the nose, rhinorrhea in particular. Slowing down of the clearance of the nasal mucosa and prolonging the contact time of locally applied drugs with the nasal mucosa would improve their efficacy. One method is creating dosage forms containing mucoadhesive polymers. We have demonstrated that a mucoadhesive solution containing HPMC enhances the clinical efficacy of oxymetazoline. However, the industrial development of fixed combinations of pharmaceutical compound and mucoadhesive carrier requires substantial investments, escalating manifold if different pharmaceutical compounds have to be rendered mucoadhesive.

NoAl is a cellulose derivative powder, which forms a gel layer on contact with the mucosal surface of the nose blocking the contact of the pollen grains with the nasal mucosa in seasonal allergic rhinitis. However, there is another potential benefit of applying NoAl (HPMC) along with other commercially available drugs for local treatment of rhinitis, as the formation of a gel layer can substantially delay their clearance from the nose and thus increase their effectiveness. This hypothesis needs to be substantiated clinically.

DETAILED DESCRIPTION:
The main objective of the trial is to test the synergy between HPMC and oxymetazoline (both applied nasally) on the increase of peak nasal inspiratory flow in patients suffering from moderately severe / severe persistent allergic rhinitis.

The design of the trial is parallel-groups, double blind, randomized, placebo controlled, single centre study.

Forty patients are randomly assigned to receive either oxymetazoline followed by HPMC (Group A) or oxymetazoline followed by placebo (Group B).

Each patient is followed up for 15 days. Day 1 is the screening and inclusion visit. Data will then be collected on day 8 & 15. Patients will fill in diaries their everyday symptoms, adverse events and applied medications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Age ≥ 18 and ≤ 50 years
* Moderately severe / severe persistent allergic rhinitis
* Positive skin prick test for perennial aero-allergens
* Active symptoms with prominent congestion at the time of inclusion

Exclusion Criteria:

* Subjects with pollen sensitization during the respective pollen season
* Subjects with arterial hypertension, arrhythmia or evidence of heart ischemia
* Subjects with other serious chronic comorbidities and bad therapeutic control
* Subjects with nasal polyposis
* Flu-like episode during the past 30 days
* Subjects unable to give informed consent
* Subjects with any of the contra-indications of oxymetazoline or NoAL
* Pregnant or lactating women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Peak nasal inspiratory flow (PNIF) area under the curve (AUC) change between the placebo and active NoAl treatment on day 1 | PNIF on Day 1, 8 and 15

SECONDARY OUTCOMES:
Difference between the PNIF AUC D1-D8 differences between the two groups | PNIF on D1 and D8
Differences in nasal mucociliary clearance (Saccharine test) between both groups. | Performed on D1, D8 and D15
Visual analogue scale (VAS) for the separate rhinitis symptoms between the two groups | On D1, D8 and D15
Change of each symptom score for congestion over 8 days | From D1 to D8
Change of total rhinitis symptom score (TRSS) over 8 days | From D1 to D8
Difference in the applied rescue decongestant (total number of additional puffs of oxymetazoline or any other medications indicated for the treatment of allergic rhinitis) as needed between the two groups | For 15 days
Number and severity of adverse events | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Todor A Popov, MD, PhD, Principal Investigator — Medical University Sofia
Locations (1):
- Medical University Sofia, University Hospital "Alexandrovska", Clinic of Allergy and Asthma, Sofia, Bulgaria

REFERENCES:
- [Background] Tzachev CT, Mandajieva M, Minkov EH, Popov TA. Comparison of the clinical efficacy of standard and mucoadhesive-based nasal decongestants. Br J Clin Pharmacol. 2002 Jan;53(1):107-9. doi: 10.1046/j.0306-5251.2001.01525.x. PMID 11849202
- [Derived] Valerieva A, Popov TA, Staevska M, Kralimarkova T, Petkova E, Valerieva E, Mustakov T, Lazarova T, Dimitrov V, Church MK. Effect of micronized cellulose powder on the efficacy of topical oxymetazoline in allergic rhinitis. Allergy Asthma Proc. 2015 Nov-Dec;36(6):e134-9. doi: 10.2500/aap.2015.36.3879. Epub 2015 Jun 29. PMID 26133030